CLINICAL TRIAL: NCT02092558
Title: Evaluation of Immunological Disorders of T Lymphocytes and Endocrinological Disorders as Pathogen Factors in Patients With Metaplasia of Urinary Bladder
Status: Completed | Type: Observational
Sponsor: Children's Hospital, Dziekanów Leśny, Poland (Other)
Responsible Party: Principal Investigator, Beata Jurkiewicz, PhD MD, Children's Hospital, Dziekanów Leśny, Poland
Other Study IDs: KB/677/09; Bioethics Commitee of Regional (Registry Identifier: KB/677/09); KB/677/09
Record Dates: First submitted 2014-03-14; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: The Follow-up Duration Was 1-8 Years.; The Main Reasons Behind Visiting the Hospital Were Recurrent Urinary Tract Infection,; Urinary Urgencies, Pollakiuria, Difficulty in Initiating Micturition, Pain in Hypogastrium,; Night Wetting and Day Wetting, Menstruation's Disorders, Urolithiasis, Defects of Urinary; System and Hematuria.
Keywords: metaplasia, dysfunction, urinary bladder, children
MeSH Terms: conditions — Urolithiasis; Hematuria; Metaplasia | interventions — Second Generation Cephalosporins; Nitrofurantoin; Cephalosporins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Female 1: Owing to the absence of an established treatment modality for squamous metaplasia of the urinary bladder in children, we developed our own treatment modalities. Children presenting with recurrent urinary tract infections on medical interview, were subjected to ultrasonography of the urinary system, repeated urinalysis, and urine culture tests. Then, on the basis of antibiogram findings, antibiotic and chemotherapeutic treatment was administered to eliminate the bacteriological factors. Second-generation cephalosporin was prescribed for 10 days, and then treatment crossover with chemotherapeutics in therapeutic dose (change in every week) during 3 months.
  Interventions: Drug: Second-generation cephalosporin, nitrofurantoin, 1% aminoglycoside solution
- Male 2: Owing to the absence of an established treatment modality for squamous metaplasia of the urinary bladder in children, we developed our own treatment modalities. Children presenting with recurrent urinary tract infections on medical interview, were subjected to ultrasonography of the urinary system, repeated urinalysis, and urine culture tests. Then, on the basis of antibiogram findings, antibiotic and chemotherapeutic treatment was administered to eliminate the bacteriological factors. Second-generation cephalosporin was prescribed for 10 days, and then treatment crossover with chemotherapeutics in therapeutic dose (change in every week) during 3 months.
  Interventions: Drug: cephalosporin with chemotherapeutics

INTERVENTIONS:
Drug: Second-generation cephalosporin, nitrofurantoin, 1% aminoglycoside solution
  Groups: Female 1
Drug: cephalosporin with chemotherapeutics — Second-generation cephalosporin was prescribed for 10 days, and then treatment crossover with chemotherapeutics in therapeutic dose (change in every week) during 3 months
  Groups: Male 2

SUMMARY:
Background: Squamous metaplasia refers to the pathological transformation of the urothelium leading to non-keratinised stratified squamous metaplasia (N-KSM).

Objective: To present the investigators experiences in the diagnosis and treatment of N-KSM of the urinary bladder in children.

DETAILED DESCRIPTION:
Design, setting, and participants: In this study, the investigators present their experiences in the diagnosis and treatment of N-KSM of the urinary bladder in children aged from 5 to 17 years. From 2005 to 2013, metaplasia was diagnosed in 119 patients - 116 girls and 3 boys. The reasons behind visiting the hospital were non-specific intense pain in the abdomen, recurrent urinary tract infections, and urination disorders. The most common symptoms of urinary bladder dysfunction were pollakiuria and difficulties in initiating micturition and retention of urine (reduced detrusor muscle activity).

Outcome measurements and statistical analysis: In 20 patients (16.8%), metaplasia was incidentally diagnosed during cystoscopy performed for other causes. Only the children whose bladders showed metaplastic changes on cystoscopy were subjected to a bladder biopsy for collecting specimens for further histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* The follow-up duration was 1-8 years.
* The main reasons behind visiting the hospital were:

  1. recurrent urinary tract infection,
  2. urinary urgencies,
  3. pollakiuria,
  4. difficulty in initiating micturition,
  5. pain in hypogastrium,
  6. night wetting and day wetting,
  7. menstruation's disorders,
  8. urolithiasis,
  9. defects of urinary system and hematuria.

Exclusion Criteria:

* No confirmation of squamous metaplasia of the urinary bladder in diagnostic cystoscopy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In all, 119 children (116 girls and 3 boys), aged between 5 and 17 years (mean age, 13.7 years), who were treated in the Pediatric Surgery Department during the period of 2005-2013 were included in this study
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Symptoms of stratified squamous metaplasia of urinary bladder and treatment's ways | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Marii Konopnickiej Street 65, Dziekanów Lesny, Poland

REFERENCES:
- See also: Bioethics Commitee in Warsaw — http://www.oil.org.pl/xml/oil/oil68/tematy/komisje/stale/bioetyki